CLINICAL TRIAL: NCT06294938
Title: Determination of Glycemic Index of Cacao Fruit Pulp
Brief Title: Glycemic Index of Cacao Fruit Pulp in Healthy, Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mars Wrigley (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M.WRI-2023-INQ-2224
Record Dates: First submitted 2024-01-12; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Blood Sugar; High; Blood Sugar; Low
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: acute, open-labeled, randomized design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose (Active Comparator): Dextrose matched for available carbohydrate
  Interventions: Other: Dextrose
- Cacao fruit pulp (Experimental): Cacao fruit pulp matched for available carbohydrate
  Interventions: Other: Cacao fruit pulp

INTERVENTIONS:
Other: Cacao fruit pulp — Cacao pulp puree
  Arms: Cacao fruit pulp
Other: Dextrose — Dextrose beverage
  Arms: Dextrose

SUMMARY:
Cacao fruit pulp is a sweet and fruity carbohydrate-rich edible mucilage that is often discarded. The objective of this study is to assess the glycemic response and determine the glycemic index of cacao fruit pulp.

DETAILED DESCRIPTION:
In an acute, open-labeled, randomized design, individuals without diabetes were studied over 120 minutes after consuming 25 grams of available carbohydrate portions of cacao pulp or dextrose.

ELIGIBILITY:
Inclusion Criteria: Subjects were males or non-pregnant females and in good health.

Exclusion Criteria: Subjects with a known history of AIDS, hepatitis, diabetes or a heart condition. Subjects taking medication or with any condition that might make participation dangerous to the subject, to others, or affect the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose | 1-120 minutes
  Mean plasma glucose
Incremental area under the curve | 1-120 minutes
  Calculated from mean plasma glucose
Peak plasma glucose | 1-120 minutes
  Peak plasma glucose (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Onterio, Canada

IPD SHARING:
Plan to Share IPD: No